CLINICAL TRIAL: NCT06074146
Title: Long-term Outcomes After Epigastric Hernia Repair in Women - a Nationwide Database Study
Brief Title: Outcomes After Epigastric Hernia Repair in Women.
Acronym: EPI-WOMEN
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Mette Willaume, Senior registrar, Bispebjerg Hospital
Other Study IDs: EPI-WOMEN
Record Dates: First submitted 2023-08-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Epigastric Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

SUMMARY:
Nationwide cohort study on women undergoing epigastric hernia repair

DETAILED DESCRIPTION:
Women have the highest prevalence of epigastric hernia repair. Outcomes after epigastric hernia repair are rarely reported independently, although pathology and surgical techniques may be different than for other primary ventral hernias.

The aim of this study was to evaluate long-term outcomes after epigastric hernia repairs in women on a nationwide basis.

Methods Nationwide cohort study from the Danish Hernia Database. Complete data from women undergoing elective epigastric hernia repair during a 12-year period (2007-2018) was extracted. A 100% follow-up was obtained by combining data from the National Civil Register. The primary outcome was operation for recurrence, secondary outcomes were readmission and operation for complications. Outcomes for open sutured repair, open mesh repair mesh, and laparoscopic repairs were compared.

ELIGIBILITY:
Inclusion Criteria:

* females undergoing epigastric hernia repair in Denmark

Exclusion Criteria:

* emergency repair umbilical hernias incisional hernias males

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identity
Study Population: females in Denmark undergoing epigastric hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 3031 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
hernia recurrence | end of study
  reoperation for recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Mette Willaume, Copenhagen, Denmark